CLINICAL TRIAL: NCT05717686
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of AHB-137 with Single Ascending Doses and Multiple Doses in Healthy Volunteers and Initial Efficacy in Chronic Hepatitis B Patients
Brief Title: A Study Evaluating AHB-137 in Healthy Participants and Participants with Chronic Hepatitis B
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AusperBio Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AB-10-8001
Record Dates: First submitted 2023-01-20; First posted 2023-02-08 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part A: SAD in healthy participants (Experimental): Part A: Single ascending doses of up to 450 mg AHB-137 by subcutaneous (SC) injection in healthy participants.
  Interventions: Drug: AHB-137 injection; Drug: Placebo
- Part B: MD in healthy participants (Experimental): Part B: Multiple doses of 300 mg AHB-137 by subcutaneous (SC) injection in healthy participants.
  Interventions: Drug: AHB-137 injection; Drug: Placebo
- Part C: MD in CHB patients (open label) (Experimental): Part C: Multiple doses of 300 mg AHB-137 by subcutaneous (SC) injection in CHB patients.
  Interventions: Drug: AHB-137 injection
- Part D: MD in CHB patients in multiple centers (Experimental): Part D: Multiple doses of 200 mg or 300 mg AHB-137 by subcutaneous (SC) injection in CHB patients (Multiple centers across multiple regions).
  Interventions: Drug: AHB-137 injection; Drug: Placebo

INTERVENTIONS:
Drug: AHB-137 injection — AHB-137 will be administered
Drug: Placebo — Placebo will be administered
  Arms: Part A: SAD in healthy participants; Part B: MD in healthy participants; Part D: MD in CHB patients in multiple centers

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics of AHB-137 subcutaneous injection in healthy volunteers and in chronic hepatitis B (CHB) patients after single and multiple doses. In addition, the study will evaluate the initial antiviral efficacy of AHB-137 in CHB patients following a multiple dosing regimen.

DETAILED DESCRIPTION:
This is a first-in-human study of AHB-137, consisting of four parts. Parts A and B are randomized, double-blinded, placebo-controlled studies designed to assess the safety, tolerability, pharmacokinetics of AHB-137 following subcutaneous injection in healthy volunteers at a 6:2 ratio of AHB-137 to placebo. Part A is a single-ascending dose (SAD) study, and Part B is a single-ascending dose (SAD) study, and Part B is a multiple dose (MD) study. Part C is an open label MD study with up to 6 CHB patients. Part D is a double blinded study in CHB patients at a 4:1 ratio to receive AHB-137 or placebo.

Study advancement to subsequent parts/cohorts will require satisfactory interim reviews of available cumulative safety data by the Safety Review Committees (SRC), using the safety criteria and review procedures described in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants are required to meet all the following inclusion criteria in order to be enrolled in the study:

  1. 18-65 years old male or female.
  2. Body Mass Index (BMI) between 19 to 35 kg/m2 (inclusive) and body weight equal to or over 45 kg.
  3. Participants' COVID-19 PCR test should be negative during screening.
  4. Participants' COVID-19 Rapid Antigen Test (RAT) should be negative at check-in.
* CHB patients are required to meet all the following inclusion criteria in order to be enrolled in the study:

  1. Have given written informed consent (signed and dated) and any authorizations required by local law and is able to comply with all study requirements.
  2. Age 18 to 65 years old.
  3. ALT ≤ 5 ULN for CHB patients recruited to Part C; ALT ≤ 2 ULN for CHB patients recruited to Part D.
  4. CHB patients who have documented chronic HBV infection equal to or above 6 months prior to screening. Otherwise, CHB patients need to be HBsAg positive and IgM HBcAb negative.
  5. CHB patients participating in Part D should have been on commercially available HBV OAV treatment(s) for at least 6 months with no change in regimen for 3 months prior to screening. HBV DNA under limit of quantification (LOQ) at Screening.
  6. Both HBeAg positive and negative CHB patients can be recruited to Part C of the study. Only HBeAg negative CHB patients can be recruited to Part D of the study.
  7. COVID-19 RAT test should be negative at check-in.

Exclusion Criteria:

* Healthy participants are required to not meet any of the following exclusion criteria in order to be enrolled in the study:

  1. Pregnant (positive pregnancy test) or lactating women. Male participants without using proper contraceptives (e.g. condom) with partners who are pregnant or lactating.
  2. History or symptoms of any clinically significant gastrointestinal, renal, hepatic, bronchopulmonary, neurological, psychiatric, cardio-vascular, endocrinological, hematological or allergic disease, metabolic disorder, cancer or cirrhosis.
  3. Personal history of congenital long QT syndrome or family history of sudden cardiac death.
  4. Any confirmed significant allergic reactions (urticaria or anaphylaxis) against any drug, or multiple drug allergies (non-active hay fever is acceptable).
  5. Any clinically significant concomitant diseases or condition that could interfere with, or treatment of which might interfere with, the conduct of the study, or that would, in the opinion of the Investigator, pose an unacceptable risk to the participant in this study.
  6. Clinically relevant electrocardiogram (ECG) abnormalities on screening ECG.
  7. ECG with QRS and/or T-wave judged to be unfavorable for a consistently accurate QT measurement.
  8. Creatinine clearance (CrCl) cutoff ≤ 60 ml/min (using the Cockcroft-Gault formula).
  9. Positive test at screening of any of the following: hepatitis A (HAV IgM Ab), hepatitis B (HBsAg), hepatitis C (HCV RNA or HCV Ab), human immunodeficiency virus 1 and 2 (HIV Ab), or TP-Ab.
  10. Any other clinically significant abnormalities in laboratory test results at screening. In the case of uncertain or questionable results, tests performed during screening may be repeated before randomization to confirm eligibility.
  11. History of bleeding diathesis or coagulopathy.

CHB patients are required to not meet any of the following exclusion criteria in order to be enrolled in the study:

1. History of liver cirrhosis and/or evidence of cirrhosis as determined by any 1 of the following:

   1. Liver biopsy (i.e., Metavir Score F4) within 2 years of screening, or
   2. FibroScan > 12 KPa, within 12 months of screening, or
   3. AST-to-Platelet Index (APRI) > 2 and FibroSure result > 0.7 within 12 months of screening.

   For patients without a test for cirrhosis in the above timeframes, FibroScan, or APRI and FibroSure, may be performed during the screening period to rule out cirrhosis History of liver failure as evidenced by ascites, hepatic encephalopathy, and/or gastric or esophageal varices.
2. History of liver disease other than hepatitis B.
3. Co-infection with TP, HCV, HIV, or hepatitis D virus (HDV).
4. Body mass index >35 kg/m2 .
5. History or suspected presence of vasculitis .
6. Diagnosed hepatocellular carcinoma or suspected hepatocellular carcinoma as evidenced by screening alpha-fetoprotein ≥200 ng/mL. If the screening alpha-fetoprotein is ≥50 ng/mL and <200 ng/mL, the absence of liver mass must be documented by imaging within 6 months before randomization.
7. Clinically relevant electrocardiogram (ECG) abnormalities on screening ECG.
8. Screening laboratory results as follows, or any other clinically significant abnormalities in screening laboratory values that would render a patient unsuitable for inclusion.

   1. ALT > 5 x ULN for Part C or > 2 x ULN for Part D
   2. Total bilirubin > 1.25 x ULN
   3. Serum albumin < 3.4 g/dL
   4. International normalized ratio of prothrombin time > 1.25
   5. Platelet count <140 x 10^9/L
   6. Hemoglobin <12.0 g/dL for males and <11.0 g/dL for females
   7. White blood cell count <3.0 k/mm3
   8. Serum creatinine >1.1 x ULN
   9. Urine protein/creatinine ratio ≥0.2 mg/mg. In the event of a ratio above this threshold, eligibility may be confirmed by a quantitative total urine protein measurement of <150 mg/24 hour
   10. Positive test (including trace) for blood on urinalysis. In the event of a positive test, eligibility may be confirmed with urine microscopy showing <5 red blood cells per high power field
9. Clinically significant abnormalities and/or poorly controlled medical conditions (e.g. Cardiovascular, pulmonary, metabolic disease) in the opinion of the investigator.
10. History of bleeding diathesis or coagulopathy.
11. History of extrahepatic disorders possibly related to HBV immune complexes (e.g., glomerulonephritis, polyarteritis nodosa) .
12. Active infection other than HBV, requiring systemic antiviral or antimicrobial therapy that will not be completed prior to Study Day 1.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2025-01-07 (Actual)

PRIMARY OUTCOMES:
Proportion of Participants With Treatment-Emergent Adverse Events (TEAEs) in Healthy Volunteers | Up to 30 days for SAD, up to 113 days for MD
Proportion of Participants With Treatment-Emergent Adverse Events (TEAEs) in CHB patients | Up to 204 days for MD

SECONDARY OUTCOMES:
The anti-HBV efficacy of AHB-137: evaluate the change in serum HBsAg (log10 IU/mL) from baseline. | Up to 204 days
The anti-HBV efficacy of AHB-137: evaluate the expression of HBsAb in serum. | Up to 204 days
The pharmacokinetic profile of AHB-137: the maximum observed plasma concentration (Cmax) of AHB-137 | Up to 30 days for SAD; up to 204 days for MD
The pharmacokinetic profile of AHB-137: time of observed maximal concentration (Tmax) of AHB-137 | Up to 30 days for SAD; up to 204 days for MD
The pharmacokinetic profile of AHB-137: areas under the concentration time curve (AUC) of AHB-137 | Up to 30 days for SAD; up to 204 days for MD
The pharmacokinetic profile of AHB-137: mean residence time (MRT) of AHB-137 | Up to 30 days for SAD; up to 204 days for MD
The pharmacokinetic profile of AHB-137: terminal half-life (t1/2) of AHB-137 | Up to 30 days for SAD; up to 204 days for MD
The pharmacokinetic profile of AHB-137: apparent subcutaneous plasma clearance (CL/F) of AHB-137 | Up to 30 days for SAD; up to 204 days for MD
The pharmacokinetic profile of AHB-137: amount of AHB-137 excreted in urine (Ae) | Day 1-4 for SAD; Day 1-4 and Day 22-25 for MD
The pharmacokinetic profile of AHB-137: renal clearance (CLr) of AHB-137 | Day 1-4 for SAD; Day 1-4 and Day 22-25 for MD

CONTACTS AND LOCATIONS:
Overall Officials: Ed Gane, Principal Investigator — University of Auckland, New Zealand
Locations (9):
- United States (4):
  - Stanford Medicine, Redwood City, California
  - University of Maryland Baltimore, Baltimore, Maryland
  - NYU Langone Health, New York, New York
  - American Research Corporation, Houston, Texas
- Queen Mary Hospital, Hong Kong, Hong Kong
- New Zealand Clinical Research, Grafton, Auckland, New Zealand
- Taiwan (3):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung, Taiwan
  - E-DA Hospital, Kaohsiung, Taiwan
  - Chia-Yi Christian Hospital, Chiayi City

IPD SHARING:
Plan to Share IPD: No